CLINICAL TRIAL: NCT03676088
Title: Comparative Evaluation of rhPDGF- BB With Modified Coronally Advanced Tunnel and CTG Versus Modified Coronally Advanced Tunnel With CTG Alone for Root Coverage in Multiple Mandibular Gingival Recession Defects- A RCT
Brief Title: Comparative Evaluation of CTG With and Without rhPDGF- BB Using Modified Coronally Advanced Tunnel for Root Coverage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02_D012_71663
Record Dates: First submitted 2018-05-08; First posted 2018-09-18 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: The patients were assigned into two treatment groups (test and control). The test group was treated with recombinant human Platelet Derived Growth Factor-BB and Modified Coronally Advanced Tunnel +Connective Tissue Graft whereas the control group was treated by Modified Coronally Advanced Tunnel +Connective Tissue Graft alone.
Who Masked: Outcomes Assessor
Masking Description: Computer generated randomization sequence was obtained by the assistant. Allocation concealment was achieved using a sealed coded opaque envelope containing the treatment of the specific subject The sealed envelope containing treatment assignment was opened immediately prior to surgery to prevent surgeon bias
Oversight: FDA-regulated Drug: No

ARMS (2):
- Test group - rhPDGF-BB+MCAT+CTG (Experimental): Root coverage surgical procedure.The patients were assigned into two treatment groups (test and control). Intervention - The test group recession coverage is treated with modified coronally advanced tunnel with connective tissue graft with recombinant human platelet derived growth factor- BB
  Interventions: Procedure: root coverage
- Control group - MCAT+CTG (Active Comparator): Root coverage surgical procedure.The patients were assigned into two treatment groups (test and control). Intervention - The control group recession coverage is treated with modified coronally advanced tunnel with connective tissue graft alone
  Interventions: Procedure: root coverage

INTERVENTIONS:
Procedure: root coverage — recession coverage is treated with modified coronally advanced tunnel with connective tissue graft with recombinant human platelet derived growth factor- BB for Experimental: Test group and without recombinant human platelet derived growth factor- BB for Active Comparator: Control group
  Other Names: root coverage with/without growth factor

SUMMARY:
The present study is a human, prospective, single centre, single blind, comparative controlled randomized clinical trial for the treatment of Miller's Class I, II or combination of class I and II mandibular recession and comparing the clinical outcomes prior to and 6 months after treatment. The trial is in accordance to the Consolidated Standards of Reporting Trials (CONSORT) criteria, 2010.

DETAILED DESCRIPTION:
24 recession defects were selected in patients who were systemically and periodontally healthy, satisfying the determined inclusion criteria. Patients with at least two or more teeth having Miller's class I , II or combination of class I and II mandibular recession defects were included in the study. A detailed, thorough medical and dental history was obtained and each patient was subjected to comprehensive clinical and radiological examination. All patients were informed about the nature of the study, surgical procedure involved, potential benefits and risks associated with the surgical procedure and a written informed consent was obtained from all patients.

The patients were assigned into two treatment groups (test and control). The test group was treated with recombinant human Platelet Derived Growth Factor-BB and Modified Coronally Advanced Tunnel +Connective Tissue Graft whereas the control group was treated by Modified Coronally Advanced Tunnel +Connective Tissue Graft alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the following criteria were included in the study:-

  * Two or more teeth with Miller's class I and II or combined class I and II recession defects in mandibular anteriors.
  * Age group 21-58 years.
  * Patients with healthy or treated periodontal conditions.
  * Patients willing to participate in the study.
  * Absence of uncontrolled medical conditions.
  * Patients with full mouth plaque score </= 10%(O'Leary 1972)
  * Patients with esthetic concerns.
  * Patients with thick gingival biotype >0.8mm

Exclusion Criteria:

* Pregnant or lactating females.
* Tobacco smoking.
* Uncontrolled medical conditions.
* Untreated periodontal conditions.
* Use of systemic antibiotics in the past 3 months.
* Patients treated with any medication known to cause gingival hyperplasia.
* Drug and alcohol abuse
* No occlusal interferences.
* Patient with a known hypersensitivity to rhPDGF-BB.

Ages: 21 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Gingival recession depth (GRD) | 6 months
  measured as the distance from the Cemento Enamel Junction to the gingival margin
2. Gingival Recession Width (GRW) | 6 months
  measured as the distance between the mesial gingival margin and distal gingival margin
Mean root coverage(MRC) | 6 months
  (Baseline recession depth - 6 month recession depth/Baseline recession depth)*100
Complete root coverage(CRC) | 6 months
  root coverage regarded as complete with gingival margin located at the level of Cemento Enamel Junction
coverage esthetic score(RCES) | 6 months
  The Aesthetic evaluation was performed according to the root coverage aesthetic score system (RES)
  Five Variables evaluated which are as follows:
  1. Level of Gingival margin (GM)
  2. Marginal Tissue Contour (MTC)
  3. Soft Tissue Texture (STT)
  4. Mucogingival Junction(MJ) alignment
  5. Gingival Colour (GC)

SECONDARY OUTCOMES:
probing pocket depth (PD) | 6 months
  measured as the distance from the gingival margin to the base of gingival sulcus
clinical attachment level (CAL) | 6 months
  measured as Gingival Recession Depth + Probing Depth
width of keratinized tissue (KTW) | 6 months
  measured as the distance from the mucogingival junction to the gingival margin , with the mucogingival junction location determined using a visual method (Schiller's Potassium Iodide Solution).

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Joann P George, MDS, Study Director — Krishnadevaraya College of Dental Sciences

IPD SHARING:
Plan to Share IPD: No